CLINICAL TRIAL: NCT03984123
Title: The Acute and Chronic Effects of Remote Ischemic Conditioning on Endothelial Glycocalyx Integrity, Cardiovascular Function and Biomarkers
Brief Title: The Acute and Chronic Effects of Remote Ischemic Conditioning on Cardiovascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate Professor of Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 301/27-6-14
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Remote Ischemic Conditioning; Endothelial glycocalyx; Arterial stiffness; micro RNA; NO pathway

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Double cuff inflation (Other): The first arm utilizes two ischemic stimuli by brachial cuff inflation of both arms at 200 mmHg for 5 minutes, separated by 15 minutes, after a baseline vascular function assessment (T0). Each ischemic stimulus is followed by a vascular function assessment (T1, T2), with a final assessment 25 minutes after the second cuff deflation (T3). All measurements are preceded by a sham conditioning procedure, by way of cuff inflation omission after their placement around the ordinary brachial position. Blood samples are drawn at baseline (T0) and at the termination of each protocol (T3). Follow-up echocardigraphy is perfomed at 1 and 2 years after inclusion to assess remodelling of left ventricle by measurmemet of left ventricular end-systolic and end-diastolic volume of left ventricle
  Interventions: Device: Brachial cuff, in order to achieve ischemic stimuli
- Single cuff inflation (Other): The second arm utilizes two ischemic stimuli by brachial cuff inflation of both arms at 200 mmHg for 5 minutes, separated by 15 minutes, after a baseline vascular function assessment (T0). Each ischemic stimulus is followed by a vascular function assessment (T1, T2), with a final assessment 25 minutes after the second cuff deflation (T3). All measurements are preceded by a sham conditioning procedure, by way of cuff inflation omission after their placement around the ordinary brachial position. Blood samples are drawn at baseline (T0) and at the termination of each protocol (T3). Follow-up echocardigraphy is perfomed at 1 and 2 years after inclusion to assess remodelling of left ventricle by measurmemet of left ventricular end-systolic and end diastolic volume of left ventricle
  Interventions: Device: Brachial cuff, in order to achieve ischemic stimuli
- Standard treatment (No Intervention): The third arm utilizes no cuff inflation to cause remote conditioning and serves as control group. Follow up echocardiography is perfomed at 1 and 2 years after inclusion to assess remodelling of left ventricle by measurmemet of left ventricular end-systolic and end diastolic volume of left ventricle

INTERVENTIONS:
Device: Brachial cuff, in order to achieve ischemic stimuli — Standard treatment with no brachial cuff inflation
  Other Names: Standard treatment
  Arms: Double cuff inflation; Single cuff inflation

SUMMARY:
The investigators are going to examine 270 patients within 48h of STEMI with primary percutaneuous intervention. The investigators utilise either a double -with a 15- min intervening interval-, or a single ischemic stimulus by brachial cuff inflation of both arms at 200mmHg for 5 min to cause remote conditioning (RIC) or no cuff inflation. Each ischemic stimulus is followed by a vascular function assessment, with a final assessment 25 minutes after the second cuff deflation. All patients utilising a cuff inflation procedure also undergo a sham cuff inflation. The investigators measure: a) the perfusion boundary region (PBR-micrometers) of the sublingual arterial microvessels as a marker of endothelial glycocalyx thickness to assess vascular permeability, b) the carotid-femoral pulse wave velocity (PWV). At baseline (T0) and the last vascular assessment (T3) The researchers also measure microRNA-144,-150,-499 (cardioprotective action), -21, and -208 (remodeling stimuli) expression, nitrate- nitrite (NOx) and malondialdehyde (MDA) plasma levels. Moreover, the investigators are going to perform an echocardiographic study at 1 and 2 years after the recruitment to investigate whether the left ventricular function differs among the 3 study arms (2 RIC protocols and no intervention)

DETAILED DESCRIPTION:
The present study is a prospective, randomized trial conducted at the Second University Department of Cardiology in Attikon University Hospital. A two hundred seventy patients with STEMI , within 48 hours after primary PCI are randomized in two remote conditioning (RIC) protocols or no intervention other than standard treatment (control group). The first protocol utilizes two ischemic stimuli by brachial cuff inflation of both arms at 200 mmHg for 5 minutes, separated by 15 minutes, after a baseline vascular function assessment (T0). Each ischemic stimulus is followed by a vascular function assessment (T1, T2), with a final assessment 25 minutes after the second cuff deflation (T3). The second protocol is identical with the first, except for the omission of the second ischemic stimulus. Both protocols are preceded by a sham conditioning procedure, by way of cuff inflation omission after their placement around the ordinary brachial position. The RIC protocol will be also performed in 30 healthy volunteers. Blood samples are drawn at baseline (T0) and at the termination of each protocol (T3). All patients are in sinus rhythm, while exclusion criteria include Killip class>2 during the index event, administration of nitrates, history of previous known coronary artery or other cardiovascular disease, previous PCI or coronary artery bypass surgery (CABG), as well chronic inflammatory and systemic disease. Furthermore, The investigators are going to conduct a two - year follow up in order to asess a) changes in left ventricular contractility via estimation of Left Ventricular End Systolic Volume( LVESV) by echocardiography study b) changes in endothelial glycocalyx and arterial stiffness.

Arterial stiffness is assessed by carotid-femoral pulse wave velocity (PWV) using arterial tonometry (Complior, Alam Medical, Vincennes, France); normal values <10 m/s. PWV is calculated as the distance between the carotid and femoral arterial pulse palpation site, divided by the transit time between waves (m/s). All measurements are performed by the same examiner, who is blind to the ischemic protocol exploited (intra-observer variability=5%).

The perfusion boundary region (PBR) of sublingual arterial microvasculature (diameter span from 5 to 25 μm) is measured using Sidestream Darkfield imaging (Microscan, Glycocheck, Microvascular Health Solutions Inc., Salt Lake City, UT, USA). The PBR is the cell-poor layer, resulting from the phase separation between the flowing red blood cells (RBC) and plasma on the microvessel luminal surface. The PBR includes the component of glycocalyx that does allow cell penetration. Thus, an increased perfused boundary region (PBR) is consistent with deeper penetration of erythrocytes into glycocalyx, indicating a loss of glycocalyx barrier properties and is a marker of reduced glycocalyx thickness. This constitutes a standardized, reproducible, operator-independent method of assessing arterial glycocalyx, and is thus proposed as a means to endothelial integrity evaluation.

Malondialdehyde (MDA) is determined spectrophotometrically with a commercial kit (Oxford Biomedical Research, Rochester Hills, Mich, colorimetric assay for lipid peroxidation; measurement range 1-20 nmol/L; 3.39% and 4.75% intra-assay and inter-assay variability respectively). IL-6 is measured by a high-sensitivity immunoassay [human IL-6 Quantikinine (high sensitivity)], that detects values as low as 0.094 (intra-assay variability <5%).

MicroRNAs (Mirs) are small, single stranded, non-coding RNA molecules comprising 19-25 nucleotides that regulate post-transcriptional gene expression in response to cellular or environmental stimuli [38]. Their non-invasiveness and stability in serum allows prompt estimation of their expression using archived serum samples. Specific MiRs have been implicated in the pathogenesis of cardiovascular disease and IRI. MiR-144 serves as a pivotal RIC mediator, while miR-150 and miR-499 inhibit apoptosis and fibrosis in the setting of animal models of myocardial IRI [40, 41]. In addition, miR-21 has been demonstrated to reduce infarct size and early left ventricular (LV) remodelling after IRI in rats. On the contrary, miR-208 exerts deleterious effects by way of hypertrophy and adverse remodelling induction . Serum miRNA are obtained from samples using the NucleoSpin miRNA Plasma Kit (MACHEREY-NAGEL GmbH & Co. KG, Duren, Germany) according to instructions of the manufacturer. The expression patterns of the miRNAs tested and a housekeeping gene, U6sn, were quantitatively assayed using reverse transcription and real-time reverse transcriptase polymerase chain reaction (RT-PCR). Stem-loop complementary DNAs (cDNAs) are synthesized using looped reverse transcription primers specific for each miRNA. Reverse transcription and quantification is performed with the Mir-X™ MicroRNA Quantification Kit (Clontech Laboratories, USA) according to the instruction of the manufacturer using Roche Light Cycler Fluorescence Quantitative PCR System (ABI, USA). All the samples are amplified in triplicate and each experiment was repeated three times to confirm reproducibility. The fold change in expression level is calculated using the 2-ΔΔCt method. The primers for PCR are:

Name Sequence miR-150 F: 5'-TCTCCCAACCCTTGTACCAGT- 3' R: 5'-GTGCAGGGTCCGAGGT-3' miR-208 F: 5'-CTTTTGGCCCGGGTTATAC-3' R: 5'-CTGACATCCTCTAGGCTGG-3' miR-144 F: 5'-GGGGGTACAGTATAGATGAT-3' R: 5'-TGCGTGTCGTGGAGTC-3' miR-499 F: 5'-CAAAGTCTTCACTTCCCTGCCA-3' R: 5'-GATGTTTAACTCCTCTCCACGTGATC-3' miR-21 F: 5'-CCCGCCTAGCTTATCAGACTG-3' R: 5'-GCCGTCGGTGTCAACATCA-3' miR-145 F: 5'-GGCGTCCAGTTTTCCCAG-3' R: 5'-CAGTGCTGGGTCCGAGTGA-3' U6sn F: 5'-CTCGCTTCGGCAGCACA-3' R: 5'-AACGCTTCACGAATTTGCGT-3' Once considered as inert by-products of NO metabolism, nitrate (NO¬3-) and nitrite (NO2-) have recently been shown to function as recycling substrates in a process of NO regeneration , which is independent of the classic L-arginine-NO-synthase (NOS) pathway. This is of particular importance in the setting of myocardial ischemia, as the latter cascade is progressively deactivated in hypoxic environments. Thus, the nitrate-nitrite (NOx) pool should be perceived as a reservoir of NO bioactivity that complements NOS in states of low-oxygen tension. The concentration of nitrate/nitrite in blood plasma is determined using Griess reaction with a commercially available kit (Cayman's Nitrate/Nitrite Colorimetric Assay Kit 780001) as we have described previously. Each plasma sample is ultrafiltered through a 10kDa molecular weight cut-off filter (Pall Nanosep® centrifugal device with Omega membrane, Sigma Aldrich: Z722065). The filters are pre-rinsed with Ultrapure water prior to ultrafiltration of the plasma. Then, 500μL of plasma is centrifuged for 30 minutes at 14.000xg at 4οC. 40μL of the filtrate are used for the determination of nitrate/nitrite , the Griess reagents are added and the absorbance of each well was measured at 540nm using the reader Infinite 200 PRO series (Tecan). The concentration of nitrate/nitrite is determined with a nitrate/nitrite standard curve respectively using Graph Pad prism version 7 (Graph Pad Software, Inc.) according to the manufacturer's instructions. The results are expressed in μmol/L.

Moreover, the investigators are going to perform an echocardiographic study at 1 and 2 years after the recruitment to investigate whether the left ventricular function differs among the 3 arms of the study (2 RIC protocols and no intervention).

STATA v.11 and SPSS v.22 are used to analyse the data. The Shapiro-Wilk test is used to examine whether the data are normally distributed, whereas the Levene test is used to examine the homoscedasticity of the data. All non-parametric variables are compared using the Wilcoxon test for comparisons between baseline and post-intervention values and are transformed into ranks for multivariate analysis. In all analyses, the researchers use two tailed tests with p<0.05. The investigators use parametric (Pearson r) and non-parametric (Spearman rho) correlation coefficients to examine cross-sectional associations. Analysis of variance (ANOVA) for clinical and biological data is performed to test the differences among groups and all non-parametric variables are transformed into ranks before entering the analysis using a previously published methodology . ANOVA (general linear model, SPSS 22, SPSS Inc, Chicago, Ill) for repeated measurements is applied for (a) measurements of the examined vascular function and biochemical markers (at T0, T1, T2, and T3 for the former and at baseline and termination of protocol for the latter) with the parameter of time used as a within-subject factor, and (b) to test differences among the 2 RIPost protocols (single- versus double-inflation) and sham procedure using a model including age, sex, BMI, dyslipidaemia, diabetes, hypertension, concomitant medical treatments, MI location, myocardial enzymes, and number of diseased coronary vessel (>70% stenosis) as covariates. The interaction between the study groups and the covariates included in the model are also examined, while the F and p values of the interaction between time of measurement of the examined markers and study groups are also calculated. The Greenhouse-Geisser correction is used when the sphericity assumption, as assessed by Mauchly's test, is not met. Post hoc comparisons are performed with Bonferroni correction. A p-value of<0.05 is considered as statistically significant. Inter- and intra-observer variabilities (%) of vascular and biochemical markers are calculated as the SD of the differences between the first and second measurements, and are expressed as a percentage of the average value in 30 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffered a STEMI within 48 hours
* Subject underwent PCI within 48 hours

Exclusion Criteria:

* Subject has known coronary artery disease or other cardiovascular disease.
* Subject has Killip class >2 during index event
* Subject received nitrates
* Subject suffers from inflammatory disease.
* Subject suffers from systematic disease

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-11-18 (Estimated)

PRIMARY OUTCOMES:
Changes of aortic stiffness among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning | Baseline,10 minutes, 25 minutes, 45 minutes
  Changes of carotid - femoral Pulse Wave Velocity among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning

SECONDARY OUTCOMES:
Changes of endothelial glycocalyx integrity among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning | Baseline,10 minutes, 25 minutes, 45 minutes
  Changes of perfusion boundary region (PBR) of sublingual arterial microvasculature (diameter span from 5 to 25 μm) among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning
Changes of oxidative stress biomarkers among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning | Baseline, 45 minutes
  Changes of malondialdehyde plamsa levels concetrations among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning
Changes of micro RNA expression among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning | Baseline, 45 minutes
  Changes of miR144, miR150, miR499, miR21, miR145, miR208a expression among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning
Changes of Nitrate-nitrite-nitric oxide plasma concetrations among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning | Baseline, 45 minutes
  Changes of Nitrate-nitrite-nitric oxide plasma concetrations among interventions arms at baseline and during the acute phase of Remote Ischemic Conditioning
Differences of left ventricular function among interventions arms at the chronic phase of Remote Ischemic Conditioning | Baseline, 2 years
  Differences of left ventricular end systolic volume among interventions arms at the chronic phase of Remote Ischemic Conditioning
Changes of aortic stiffness among interventions arms at the chronic phase of Remote Ischemic Conditioning | Baseline, 2 years
  Changes of carotid - femoral Pulse Wave Velocity among interventions arms at the chronic phase of Remote Ischemic Conditioning
Changes of endothelial glycocalyx integrity among interventions arms at the chronic phase of Remote Ischemic Conditioning | Baseline,2 years
  Changes of perfusion boundary region (PBR) of sublingual arterial microvasculature (diameter span from 5 to 25 μm) among interventions arms at the chronic phase of Remote Ischemic Conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Vlastos, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Efstathios K. Iliodromitis, MD, PhD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Derived] Pavlidis G, Tsilivarakis D, Katogiannis K, Vlastos D, Katsanos S, Katsanaki E, Thymis J, Parissis J, Lambadiari V, Ikonomidis I. Association of aortic stiffness early post myocardial infarction with left ventricular remodelling. Eur J Clin Invest. 2024 Jan;54(1):e14090. doi: 10.1111/eci.14090. Epub 2023 Sep 7. PMID 37675585
- [Derived] Ikonomidis I, Vlastos D, Andreadou I, Gazouli M, Efentakis P, Varoudi M, Makavos G, Kapelouzou A, Lekakis J, Parissis J, Katsanos S, Tsilivarakis D, Hausenloy DJ, Alexopoulos D, Cokkinos DV, Botker HE, Iliodromitis EK. Vascular conditioning prevents adverse left ventricular remodelling after acute myocardial infarction: a randomised remote conditioning study. Basic Res Cardiol. 2021 Feb 6;116(1):9. doi: 10.1007/s00395-021-00851-1. PMID 33547969